CLINICAL TRIAL: NCT07232082
Title: Assessing Local Hypothermia and Endovascular Recanalization for Acute Stroke With a Large Core Infarction-A Multicenter, Prospective, Open-label, Blinded-Endpoint, Randomized Controlled Trial
Brief Title: Assessing Local Hypothermia and Endovascular Recanalization for Acute Stroke With a Large Core Infarction
Acronym: RESCUE-LCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20250913
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Large Ischemic Core
Keywords: endovascular therapy; Hypothermia
MeSH Terms: conditions — Stroke; Hypothermia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normothermial group (Active Comparator): In the contral group, after crossing the occluded vessel segment with a microcatheter and confirming its location in the true lumen, roomtemperature saline will be extracted from the refrigerator. 50ml will be drawn within 2 minutes and then continuously infused at a rate of 10ml/min using an infusion pump. After infusion, standard thrombectomy procedures will be performed. After completion of the thrombectomy procedure (regardless of achieving 2b/3-grade reperfusion), another roomtemperature 300ml of saline will be extracted within 2 minutes and infused at a rate of 30ml/min for 10 minutes through the intermediate catheter or guiding catheter placed in the internal carotid artery.
  Interventions: Other: Control (Normal saline)
- Hypothermia group (Experimental): In the treatment group, after crossing the occluded vessel segment with a microcatheter and confirming its location in the true lumen, 4℃-saline will be extracted from the refrigerator. 50ml will be drawn within 2 minutes and then continuously infused at a rate of 10ml/min using an infusion pump. After infusion, standard thrombectomy procedures will be performed. After completion of the thrombectomy procedure (regardless of achieving 2b/3-grade reperfusion), another 300ml of saline will be extracted within 2 minutes and infused at a rate of 30ml/min for 10 minutes through the intermediate catheter or guiding catheter placed in the internal carotid artery. Post-infusion, contrast-enhanced cerebral angiography using room temperature contrast agent is generally not recommended to dilute the local temperature.
  Interventions: Other: intra-arterial local therapeutic hypothermia

INTERVENTIONS:
Other: intra-arterial local therapeutic hypothermia — In the treatment group, after crossing the occluded vessel segment with a microcatheter and confirming its location in the true lumen, 4℃-saline will be extracted from the refrigerator. 50ml will be drawn within 2 minutes and then continuously infused at a rate of 10ml/min using an infusion pump. After infusion, standard thrombectomy procedures will be performed. After completion of the thrombectomy procedure (regardless of achieving 2b/3-grade reperfusion), another 300ml of saline will be extracted within 2 minutes and infused at a rate of 30ml/min for 10 minutes through the intermediate catheter or guiding catheter placed in the internal carotid artery. Post-infusion, contrast-enhanced cerebral angiography using room temperature contrast agent is generally not recommended to dilute the local temperature.
  Arms: Hypothermia group
Other: Control (Normal saline) — In the contral group, after crossing the occluded vessel segment with a microcatheter and confirming its location in the true lumen, roomtemperature saline will be extracted from the refrigerator. 50ml will be drawn within 2 minutes and then continuously infused at a rate of 10ml/min using an infusion pump. After infusion, standard thrombectomy procedures will be performed. After completion of the thrombectomy procedure (regardless of achieving 2b/3-grade reperfusion), another roomtemperature 300ml of saline will be extracted within 2 minutes and infused at a rate of 30ml/min for 10 minutes through the intermediate catheter or guiding catheter placed in the internal carotid artery.
  Arms: Normothermial group

SUMMARY:
A multicenter, prospective, open-label, blinded-endpoint, randomized controlled trial to assess the effectiveness and safety of catheter-based focal intracranial hypothermia combined with endovascular reperfusion therapy for acute patients with a Large Core Infarction.

DETAILED DESCRIPTION:
This trial aims to assess the effectiveness and safety of catheter-based focal intracranial hypothermia combined with endovascular reperfusion therapy for patients with acute patients with a Large Core Infarction. Participants were centrally randomized in a 1:1 ratio to either endovascular thrombectomy (EVT) combined with intra-arterial cold saline infusion (IA-CSI) (hypothermia group) or EVT combined with normothermic saline infusion (normothermia group).

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria：

1. Age ≥18 years old.
2. The National Institutes of Health Stroke Scale (NIHSS) score was ≥6 points before randomization.
3. Time from symptom onset to randomization ≤24h.
4. Patients or their guardians can understand the purpose of the trial, voluntarily participate and sign a written informed consent, and are capable of receiving clinical follow-up.

Specific Neuroimaging Inclusion Criteria

1. Prior to randomization, CTA, MRA, or DSA confirmed the presence of anterior circulatory large vessel occlusion (internal carotid artery or M1segment).
2. NCCT ASPECTS value of 3 to 5 based on findings from non-contrast CT within 24 hours after stroke onset (defined as the time the patient was last known to be well), with no limitation with respect to infarct-core volume;
3. NCCT ASPECTS value of 0 to 2 based on findings from non-contrast CT within 24 hours after stroke onset and an infarct-core volume between 70 ml and 100 ml;
4. NCCT ASPECTS value greater than 5 based on findings from non-contrast CT after stroke onset and an infarct-core volume of 70 to 100 ml.

Exclusion Criteria:

1. Pre stroke mRS>1 score.
2. Multivessel Occlusion
3. Concomitant untreated intracranial aneurysms, intracranial tumors (with the exception of small meningiomas), or intracranial vascular malformations.
4. History of intracranial hemorrhage within 6 months, including parenchymal hemorrhage, intraventricular hemorrhage, or subarachnoid hemorrhage.
5. History of gastrointestinal hemorrhage, genitourinary bleeding, acute myocardial infarction (AMI), cranial trauma, or having undergone major surgical procedures within the past month.
6. The presence of active bleeding, severe anemia, coagulation dysfunction, or an uncorrected bleeding tendency (platelet count < 40,000 /μl, uncorrected INR>2.0).
7. Patients with heart function of grade 1 or above, or with a clear history of acute or chronic heart dysfunction, are at greater risk of acute heart failure or fluid perfusion intolerance as determined by clinicians.
8. Severe heart, liver, kidney disease.
9. Known allergy to contrast media or related medications.
10. Refractory hypertension uncontrolled by medication (defined as persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg).
11. glucose <2.8 mmol/L or >22.2 mmol/L；
12. Pregnancy or lactation；
13. the expected survival time is less than 12 months.
14. Participating in other clinical trials, in the investigational phase or in the follow-up phase.
15. Other conditions deemed by investigators to pose significant risks or render participation unsuitable (e.g. inability to comply due to psychiatric/cognitive/emotional disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score 0-2 at 90 days. | 90±7 days after randomization
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.

SECONDARY OUTCOMES:
Neurofunctional deficit defined as modified Rankin Scale (mRS) | 90±7 days after randomization
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
Proportion of patients with modified Rankin Score 0-1 at 90 days | 90±7 days after randomization
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.
Proportion of patients with modified Rankin Score 0-3 at 90 days. | 90±7 days after randomization
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.
Rate of symptomatic intracranial hemorrhage within 48 hours (Heidelberg Bleeding Classification) | within 48±12 hours after randomization
  Intracranial hemorrhage (ICH) was assessed with the Heidelberg Bleeding Classification within 48 hours of endovascular treatment. Intracranial hemorrhage was classified as hemorrhagic infarction or parenchymal hematoma. The sICH was defined as ICH associated with a worsening of 4 or more points on the NIHSS or resulting in death, and cerebral herniation, which were not present at baseline.
All-Cause Mortality within 90 (±7) Days Post-Randomization | 90±7 days after randomization
  The modified Rankin Scale is a graded ordinal scale that ranges between 0 and 6, where a score of 6 is assigned to indicate mortality.
Any type of intracranial hemorrhage according to Heidelberg Classification. | within 48±12 hours after randomization
  Any type of intracranial hemorrhage according to Heidelberg Classification.
Incidence rate of malignant cerebral edema within 72 (±48) hours post-randomization | 72 (±48) hours post-randomization
  Patients with MCE were defined as those with: (1) infarct lesions with obvious space-occupying mass effect with more than 50% of the MCA territory and signs of local brain swelling such as sulcal effacement and compression of the lateral ventricle and (2) midline shift of ≥5 mm at the septum pellucidum or pineal gland with obliteration of the basal cisterns

IPD SHARING:
Plan to Share IPD: No